CLINICAL TRIAL: NCT06853665
Title: A Pharmaco-Imaging Trial of Mixed Amphetamine Salts for the Treatment of ADHD in Intellectually-intact Youth With Autism Spectrum Disorder
Brief Title: The TEAM Study - Treatment Efficacy for Autism/Attention Using Mixed Amphetamine
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gagan Joshi (Other)
Collaborators: Massachusetts Institute of Technology (MIT) (Unknown)
Responsible Party: Sponsor-Investigator, Gagan Joshi, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-P-000007
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Autism; Autism Spectrum Disorder
Keywords: ADHD; Attention; Autism; Treatment; Pharmaco-imaging; Imaging; MRI; Drug Study
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autistic Disorder; Autism Spectrum Disorder | interventions — SLI381

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Mixed Amphetamine Salts (MAS) (also known as Adderall XR) (Experimental): Participants in the MAS arm will receive MAS in capsule form daily for 4 weeks . Participants will undergo neuroimaging before and after the 4-week treatment phase.
  Interventions: Drug: Adderall XR (mixed salts amphetamine)
- Placebo (Placebo Comparator): Participants in the placebo arm will receive placebo (no active ingredients) in capsule for daily for 4 weeks. Participants will undergo neuroimaging before and after the 4-week treatment phase.
  Interventions: Drug: Placebo
- Control Group (No Intervention): Typically-developing controls will undergo neuroimaging twice (4 weeks apart) and will receive no intervention during the 4-week window.

INTERVENTIONS:
Drug: Adderall XR (mixed salts amphetamine) — Capsule
  Arms: Mixed Amphetamine Salts (MAS) (also known as Adderall XR)
Drug: Placebo — Capsule
  Arms: Placebo

SUMMARY:
The investigators are conducting a 10-week brain imaging and medication study. They are doing the research to study the response of Attention-Deficit/ Hyperactivity Disorder (ADHD) in youth with Autism Spectrum Disorder (ASD) on extended-release formulation of mixed amphetamine salts (MAS) (also know as Adderall XR). The investigators also want to find out if taking MAS has any effect on the brains of children and adolescents with ADHD and ASD. This study will help researchers better understand how the use of MAS to treat ADHD effects children and adolescents with ASD. The investigators will compare MAS to a placebo. The placebo will look exactly like the MAS capsules but will contain no MAS. During this study, participants may get a placebo instead of MAS. Placebos are used in research studies to see if the study results are due to the study drug or due to other reasons.

Participants with ASD and ADHD will complete 4-weeks of treatment with the study medication or placebo. They will complete bi-weekly study visits virtually via a telemedicine platform with the study doctor and complete questionnaires. On alternating weeks, they will meet with a Massachusetts General Hospital (MGH) study team member to discuss medication adherence and potential side effects. Participants will have the option to attend all study visits in-person if participants prefer. They will also complete baseline and endpoint Magnetic Resonance (MR) scan visits at Massachusetts Institute of Technology (MIT). During the MR Scan visits, they will complete a series of tasks to measure inattention, impulsivity, reward sensitivity, decision-making, and working memory.

Participants without ADHD or ASD will complete eligibility screening with MGH. If eligible, they will be invited to baseline and endpoint MR scan visits at MIT. During the MR Scan visits, they will complete a series of tasks to measure inattention, impulsivity, reward sensitivity, decision-making, and working memory.

ELIGIBILITY:
Inclusion Criteria:

Participants with Autism Spectrum Disorder (ASD) and Attention Deficit/Hyperactivity Disorder (ADHD)

* Male or female participants between 8 and 18 years of age (inclusive).
* Participant intact communicative language, as clinically determined.
* Meet DSM-5-TR diagnoses of ADHD and ASD as established by clinical diagnostic interview.
* At least moderate current ADHD symptoms severity (Clinician-rated ADHD-RS score ≥28 and ADHD-CGI-S of ≥4)
* At least moderate current ASD symptoms severity (SRS-2 raw score ≥85 and ASD-CGI-S of ≥4).
* Participants with disruptive behavior disorders, mood and anxiety disorders will be allowed to participate in the study provided they do not meet any exclusionary criteria.
* Participant must be on a stable regimen of psychotropic treatment.
* Participants must understand the nature of the study. Participants must be deemed not to have impaired decision-making capacity and must have the capacity to provide direct informed consent. Participants must sign an IRB-approved informed consent form before initiation of any study procedures.
* Participants must have a level of understanding sufficient to communicate with the investigator and study coordinator and be willing to cooperate with all tests and examinations required by the protocol.
* Participant weight is above the 5th percentile and below the 95th percentile, per CDC child BMI categories (https://www.cdc.gov/obesity/basics/childhood-defining.html)

Typically Developing Control Participants

* Age-, sex-, & IQ-matched with ASD participants.
* No significant traits of ASD as screened by SRS-2 (raw score <60).
* No significant ADHD symptoms as screened by parent-rated ADHD-RS (score <18)
* No significant psychopathology as screened on the CBCL (Subdomain T-scores <60).
* Participant weight is above the 5th percentile and below the 95th percentile, per CDC child BMI categories (https://www.cdc.gov/obesity/basics/childhood-defining.html)

Exclusion Criteria (all participants except where noted):

* Impaired intellectual capacity as determined either by history of intellectual disability or as assessed, in ASD participants only, during the clinical evaluation and determination will be based on intact communicative language, intellectual performance, and ability to take personal care.
* Participant is unable to communicate due to delay in, or total lack of, spoken language development (grossly impaired language skills)
* Participants with a poor command of the English language and/or require an interpreter.
* Participant is unable to swallow pills (ASD participants only)
* Participants with a medical condition or treatment that will either jeopardize subject safety or affect the scientific merit of the study, including:
* Pregnant or nursing females or females with a positive Beta-HCG pregnancy test.
* Uncorrected hypothyroidism or hyperthyroidism.
* History of non-febrile seizures within last 1 month without a clear and resolved etiology.
* Diagnosis of glaucoma (ASD participants only)
* History of renal or hepatic impairment.
* Serious systemic illness
* Personal history of cardiac disease or a family history of non-geriatric cardiac disease or death (ASD only)
* Participants with known medical risk factors (e.g., known untreated hypertension, arrhythmia, premature family history of sudden death) and active symptoms that, in the investigators' opinion, place them at risk for untoward adverse effects (ASD only)
* Participants with an unstable medical condition (that requires clinical attention).
* Clinically unstable psychiatric conditions or judged to be at serious safety risk to self (suicidal risk) or others (within past 30 days).
* Participants currently (within past 30 days) experiencing significant symptom severity of major psychiatric disorders as clinically determined.
* Active symptoms of anorexia or bulimia nervosa
* History of substance use (except nicotine, recreational use of THC, or caffeine) within past 3 months
* Initiation of a new psychosocial intervention within 4 weeks prior to randomization.
* Participants treated with a psychotropic medication(s) on a dose that has not been stable for at least 4 weeks prior to study baseline.
* Participants receiving treatment with an MAOI within two weeks prior to receiving study medication.
* Participants receiving treatment with stimulant class of medication. (ASD participants on a stable treatment of non-stimulant ADHD treatment medications will be included.)
* History of non-response of ADHD symptoms to amphetamine salt as defined by being on therapeutic dose for at least 1 week. (ASD only)
* Subjects with previous poor response or poor tolerability to mixed amphetamine salts (ASD only)
* History of allergic reaction to amphetamine or dextroamphetamine (for ASD participants only)
* Investigator and his/her immediate family, defined as the investigator's spouse, parent, child, grandparent, or grandchild.
* Contraindications to MRI scanning as described in the MIT MRI Screening Checklist. Subjects can choose a security object (e.g., fidget toy, stuffed animal, or blanket) that is MRI-safe and provided by the imaging center, in the scanner to help with possible anxiety they might experience due to the scanning. Typically developing control subjects with contraindications to MRI scanning will not be eligible to participate in the trial.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 196 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2030-01-10 (Estimated); Study Completion 2030-01-10 (Estimated)

PRIMARY OUTCOMES:
Change in the clinician-rated ADHD-Rating Scale (ADHD-RS) | Baseline to Week 4 (study endpoint)
  Efficacy will be assessed by reduction in ADHD symptoms as measured by change from baseline on the clinician-rated ADHD-Rating Scale (ADHD-RS). The ADHD-RS-V is a physician-rated scale to assess the ADHD symptom severity in participants aged 5 to 17 years old. It is an 18-item rating-scale corresponding to DSM-5 diagnostic symptom criteria. Total scores range from 0-54, where higher scores indicate greater severity. The outcome reported reflects the change from baseline in ADHD-RS score and negative scores represent improvement.
Treatment Responder | Week 4 (study endpoint)
  Responders are defined as ≥30% reduction in clinician-rated ADHD-Rating Scale (ADHD-RS) and clinician-rated Clinical Global Impression-Improvement score for ADHD (ADHD-CGI-I) ≤2 OR ≥25% reduction in parent-rated ADHD-RS and clinician-rated ADHD-CGI-I score ≤2.

SECONDARY OUTCOMES:
Pre and post treatment changes in ASD core symptoms on Social Responsiveness Scale 2 (SRS-2) | Baseline to Week 4 (study endpoint)
  Change in ASD symptoms as measured by change from baseline on the Social Responsiveness Scale 2 (SRS-2) scale. The SRS-2 is a 65-item rating scale that is used to measure the severity of autism spectrum symptoms as they occur in natural settings. The SRS-2 School Age form is completed by a parent or guardian for patients ages 9-17. Total raw scores range from 0 to 195, with higher scores indicating increased symptom severity. The outcome reported reflects the change from baseline in SRS Total raw score and negative scores represent improvement.
Pre and post treatment changes in brain functioning | Baseline to Week 4 (study endpoint)
  The study's primary neuroimaging measures include pre and post-treatment changes in brain functioning using multiple neuroimaging modalities, including resting-state functional MRI to assess connectivity in key networks (default mode, salience, and frontoparietal), task-based fMRI during response inhibition tasks to evaluate activation in inhibitory control regions, and magnetic resonance spectroscopy to analyze neurometabolite concentrations. Multimodal neuroimaging techniques will help identify neural correlates of treatment response by examining changes in large-scale network connectivity patterns (default mode, salience, and frontoparietal), task-related activation in regions previously associated with attention and inhibition (right inferior frontal gyrus, subthalamic nucleus, and anterior cingulate cortex), and alterations in brain neurochemistry (glutamate, GABA, glutathione, N-acetyl aspartate).

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No